CLINICAL TRIAL: NCT04554927
Title: Impact of Web Application Support Versus Standard Management on Compliance With Adjuvant Hormone Therapy at 18 Months in Patients Treated for Breast Cancer
Acronym: WEBAPPAC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Francois Baclesse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: WEBAPPAC
Record Dates: First submitted 2020-09-14; First posted 2020-09-18 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-08

CONDITIONS: Web-application; Breast Cancer; Hormono Therapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- WEB-application (Experimental)
  Interventions: Other: WEB-Application
- Standard accompaniment (Active Comparator)
  Interventions: Other: Standard accompaniment

INTERVENTIONS:
Other: WEB-Application — The patients of the Web-application arm will be trained on the devices and the application will be installed either on their smartphone or on another support (computer, tablet).
  Arms: WEB-application
Other: Standard accompaniment — Personalized schedule of medical follow-up given to the patient
  Arms: Standard accompaniment

SUMMARY:
The investigators hypothesize that the implementation of a Web-application in patients initiating adjuvant hormone therapy for breast cancer brings a benefit on treatment adherence and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patient > 18 years old
* Breast cancer patient candidate for adjuvant hormone therapy
* Mastery of the French language
* Patient with a cell phone and an Internet connection
* Patient able to use a computer, smartphone, or tablet.
* Patient affiliated to a social security system
* Signing of informed consent prior to any specific study-related procedure

Exclusion Criteria:

* Patient who has previously received hormone therapy for cancer.
* Patient not trained in the use of the application
* Any associated medical or psychiatric condition that might compromise the patient's ability to participate in the study
* Patients with locoregional or metastatic recurrence
* Other history of cancer.
* Patient deprived of liberty, under guardianship or curatorship
* Simultaneous participation in a therapeutic clinical trial or other clinical study involving a connected tool
* Patient unable to undergo trial follow-up for geographical, social or psychopathological reasons

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 438 (Estimated)
Dates: Start 2020-09-03 (Actual); Primary Completion 2024-10-11 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Observance of hormontherapy | 18 months
  Evaluate the benefit of a web-based application on hormone therapy compliance (Morisky questionnary; answer Yes or No; 8 questions)

SECONDARY OUTCOMES:
Quality of life with self questionnaires | 18 months
  Quality of life scores according (EORTC QLQ-C30 self-questionnaires ; minimum not at all to maximum Lot; 30 questions)
Quality of life with self questionnaires | 18 months
  uality of life scores according (EORTC QLQ-BR23 self-questionnaires ; minimum not at all to maximum Lot; 23 questions)

CONTACTS AND LOCATIONS:
Locations (1):
- Centre François baclesse, Caen, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gernier F, Grellard JM, Dupont C, Castel H, Fernette M, Lahaye F, Charles RM, Leroux T, Ory C, Faveyrial A, Morel A, Emile G, Levy C, Segura C, Allouache D, Johnson A, Geffrelot J, Gunzer K, Lelaidier A, Girault G, Dubot-Poitelon C, San C, Lequesne J, Clarisse B. Impact of web application support versus standard management on adherence with adjuvant hormone therapy in patients treated for breast cancer: the WEBAPPAC study. BMC Cancer. 2023 Aug 9;23(1):736. doi: 10.1186/s12885-023-11242-1. PMID 37559004